CLINICAL TRIAL: NCT03477240
Title: A Cross-Sectional Feasibility Study of a Telephonic Questionnaire By Research Nurses For Follow-Up Of Locally Advanced Cervical Cancer Patients With Complete Response To Treatment.
Brief Title: Feasibility Study Of A Telephonic Questionnaire For Follow-Up Of Locally Advanced Cervical Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Umesh Mahantshetty, Professor Dr., Tata Memorial Hospital
Other Study IDs: TMH-1950
Record Dates: First submitted 2018-01-11; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-02

CONDITIONS: Cervical Cancer Stage IIIB; Treatment Outcome; Follow up; QUESTIONNAIRE
Keywords: Cervical Cancer; TELEPHONIC QUESTIONNAIRE; Follow up
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cross-sectional Feasibility study on all consecutive patients of locally advanced cancer of the cervix or vault treated entirely at Tata Memorial Centre with curative intent radiation or chemoradiation.

DETAILED DESCRIPTION:
Our institution registers on an average 670 cases of cancer cervix in a year and almost 75% are treated with curative intent, therefore around 500 patients a year would be treated with curative intent. Assuming that 75% of patients registered in a year would be receiving treatment at our institute, 375 patients a year would be completing treatment, of whom the investigator expect 80-85% ,i.e 300 patients to have a complete response. The list of patients who have completed radio(chemotherapy) in 2015 &2016 can be obtained from the Radiation Oncology Department records. Patients identified for a follow up visit will be telephonically contacted between one and two weeks before the planned clinic visit and verbal telephonic consent taken prior to the nurse-led interview. This study should be able to accrue 300 patients in 6 months.

Patients of locally advanced cervical cancer or vault cancer who have been treated with radiotherapy with or without concurrent chemotherapy and have a clinical complete response at 3 months post treatment and are within the first 2 years post treatment completion will be eligible to participate in this study.

Screening: Patients will be screened from the list of patients treated in the radiotherapy department over the last 2 years (2015-2016), available from the Radiation Oncology Information System (ROIS). All patients with a diagnosis of cervical cancer or vault cancer will be screened using the hospital Electronic Medical Record (EMR) to check stage of disease, schedule of treatment received, response at 3 months post treatment and expected date of next follow up.

If patient fulfils all inclusion criteria, she will be called by the research nurse, approximately 1-2 weeks prior to her expected date of follow up, for a preliminary conversation and invited to participate in the study.

After verbal telephonic consent is obtained, she will be interviewed by the clinical research nurse using the format of the prepared proforma (Form A) regarding symptoms suggestive of disease recurrence as well as treatment induced toxicity. At the end of the interview, the research nurse records her impression of whether the patient has worrisome symptoms of disease or not and has symptoms of treatment toxicity or not for which she should visit the hospital.

When the patient reports to the OPD the next week for scheduled physical follow up, the nurse completes the consenting process by taking a short written informed consent. The examining physician then takes a complete history and in addition, performs a physical examination and any investigations he/she deems necessary. Following this he/she notes down final impression of disease status and toxicity which are taken as the gold standard (Form B). Each patient will be interviewed only once during their follow up schedule.

In addition at the physical visit, information regarding the acceptability of nurse-led telephonic follow-up to the patient and the financial impact of physical follow- up will be collected using a structured format (Form C).

Study participant drop-out/ Lost-to-follow up: Patients may withdraw their consent at any point during the telephonic interview or the subsequent follow up visit.

* A patient who does not attend the scheduled follow up visit within 1-2 weeks of the telephonic interview will be called a second time to remind her of the follow up appointment and enquire about reasons for non-attendance in the clinic, which will be recorded. If patient does not report to the clinic within the next 2 weeks, she will be considered to have dropped out from the study.
* Those patients in whom the interval between telephonic interview and the physician's assessment is more than 4 weeks, will be considered drop outs and follow up telephone call will go out to enquire about reasons for non-attendance in the clinic, which will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Cervical Cancer Stage Ib2, II and III (Squamous carcinoma or adenocarcinoma)
2. Cancer of the vault
3. Cancer of the cervix which inadvertently underwent hysterectomy (inadequate surgery)
4. Treated with curative intent with radical radio(chemo)therapy or NACT followed by radical radio(chemo)therapy and completed all curative treatment.
5. Within 2 years post completion of treatment
6. Has complete clinical response at 3 months post treatment
7. Informed consent
8. Contactable by telephone

Exclusion Criteria:

1. Patients with Stage III disease treated with palliative intent with once monthly radiotherapy
2. Early stage cervical cancer patients who underwent Wertheims hysterectomy and who have completed adjuvant radiochemotherapy due to high-risk factors
3. Metastatic cervical cancers
4. Patients who are unable to comprehend the questions or dialogue over telephone by medical staff.
5. Patients who seem unreliable for follow up

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients of locally advanced cancer of the cervix or vault treated entirely at Tata Memorial Centre with curative intent radiation or chemoradiation.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of nurse-led telephonic interview for disease recurrence | 1 YEAR
  To estimate the accuracy of nurse-led telephonic interview in identifying patients with symptoms suggestive of disease recurrence, in terms of sensitivity and specificity values

SECONDARY OUTCOMES:
Accuracy of nurse-led telephonic interview for late toxicity of treatment | 1 YEAR
  To estimate the accuracy of nurse-led telephonic interview in identifying patients with symptoms suggestive of late toxicity of treatment
Acceptability of a nurse-led telephonic surveillance program using structured format (Form C). | 1 YEAR
  To assess patients' acceptability of a nurse-led telephonic surveillance program (if found to be concordant with physical clinic visits)

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared